CLINICAL TRIAL: NCT04522466
Title: Evaluation of the Pharmacokinetics and Pharmacodynamics of Hydroxychloroquine in COVID-19 Intensive Care Unit Patients
Acronym: PREAVIS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Stop of the study by competent authority (ANSM)
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: CHU Saint-Etienne - Laboratoire de Pharmacologie - Toxicologie - Gaz du sang (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20CH065; 2020-001281-11 (EudraCT Number)
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Sars-CoV2
Keywords: SARS-CoV-2; Hydroxychloroquine; COVID-19; Intensive care unit; Pharmacokinetics
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients infected by SARS-CoV-2 treated by Hydroxychloroquine (Experimental): Blood sample on patients infected by SARS-CoV-2 treated by Hydroxychloroquine
  Interventions: Drug: Hydroxychloroquine (HCQ)

INTERVENTIONS:
Drug: Hydroxychloroquine (HCQ) — Hydroxychloroquine (HCQ) will be administered as usual practice: dosage is adjusted to maintain a concentration between 1 and 2 mg/L.
  Measure pharmacokinetics and pharmacodynamics of Hydroxychloroquine (HCQ).

SUMMARY:
To date, no treatment has demonstrated clinical efficacy on COVID 19. However, several therapeutic strategies are being considered and are being evaluated in numerous clinical trials. Among these strategies, the use of hydroxychloroquine (HCQ) seems promising. There is very little information on how to precisely administer hydroxychloroquine to patients infected with SARS-CoV-2 in intensive care, which may be responsible for side effects, some of which are potentially serious. In addition, this treatment has a long half-life which increases the risk of accumulation and therefore toxicity. In view of the lack of knowledge on the pharmacokinetic / pharmacodynamic properties of hydroxychloroquine in intensive care patients infected with SARS-CoV-2, we propose to perform a prospective multicenter cohort study in order to collect the biological data necessary for this evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years of age and older
* Patients hospitalized in the intensive care unit infected with CoV-2-SARS for whom a diagnosis of respiratory CoV-2-SARS infection has been made by nasopharyngeal swab or deep respiratory sampling.
* Patient receiving HCQ treatment as part of care or as part of a clinical trial.
* Patient affiliated or entitled to a social security scheme

Exclusion Criteria:

* Hypersensitivity to the active substances or to any of the following excipients: lactose monohydrate, povidone, corn starch, magnesium stearate.
* Retinopathies
* Combination with citalopram, escitalopram, hydroxyzine, domperidone and piperazine due to increased risk of ventricular rhythm disturbances, including torsades de pointes.
* Patient with known QT prolongation
* Known deficit in G6PD
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of hydroxychloroquine (HCQ) | Up to day 21
  measured blood concentration by blood sample results.

SECONDARY OUTCOMES:
Correlation between hydroxychloroquine (HCQ) concentration and cardiac toxicity (QT interval) | Up to day 21
  measured by blood sample and electrocardiogram results.
Correlation between Pharmacokinetic (concentration) and pharmacodynamic (viral load) of hydroxychloroquine (HCQ) | Day 1, Day 3, Day 5, Day 7, Day 14, Day 21
  measured by blood sample
Pharmacokinetic model | Up to day 21
  Pharmacokinetic (area under the curve) analysis will be performed using a population approach with a non-linear mixed effects model.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie PERINEL, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (4):
- France (4):
  - Groupement Hospitalier des Portes de Province, Montélimar
  - Centre Hospitalier de Roanne, Roanne
  - CHU Saint-Etienne, Saint-Etienne
  - Clinique Mutualiste, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No